CLINICAL TRIAL: NCT00808002
Title: Efficacy of Treatment Intensification With Maraviroc on HIV-1 Viral Latency in Recently Infected Hiv-1 naïve Patients Starting Raltegravir Plus Tenofovir/Emtricitabine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Dr . BONAVENTURA CLOTET, Dr. Bonaventura Clotet, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARAVIBOOST
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: HIV Infections
Keywords: Maraviroc; CCR5 antagonists; Primary HIV Infection; HIV-1 reservoir; eradication; treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Maraviroc; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): From Baseline to Week48: Raltegravir BID + Tenofovir/Emtricitabine QD + Maraviroc BID From W48 to W72: Raltegravir BID + Tenofovir/Emtricitabine QD
  Interventions: Drug: Raltegravir; Drug: Maraviroc; Drug: Tenofovir/Emtricitabine
- 2 (Active Comparator): Start ARV treatment with : Raltegravir BID + Tenofovir/Emtricitabine
  Interventions: Drug: Raltegravir; Drug: Tenofovir/Emtricitabine

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg every 12 hours
Drug: Maraviroc — Maraviroc 300 mg every 12 hours
  Arms: 1
Drug: Tenofovir/Emtricitabine — Tenofovir/Emtricitabine 300/200 mg every 24 hours

SUMMARY:
The intensification with maraviroc in recently HIV-1-infected patients of a preferred gold-standard triple therapy composed of raltegravir plus tenofovir/emtricitabine could accelerate the decay of the HIV-1 reservoir in latently infected cells established early in HIV-1 infection.

This could provide further insight into this area, decrease the size of latent reservoir, and translate into clinical benefits for patients.

DETAILED DESCRIPTION:
A reservoir of latently infected cells established early in infection may be involved in the maintenance of viral persistence despite continuous highly active antiretroviral therapy (HAART). This is likely to represent the major barrier to virus eradication in patients on successful combination antiretroviral therapy.

The majority of the viruses in the latent reservoir use CCR5 receptor during entry.

More recently, clear evidences for decay of this HIV-1 reservoir in patients who initiated antiretroviral therapy early in infection have been demonstrated. The treatment of acute infection may set the stage for subsequent attempts at eradication. To achieve this, more potent antiretroviral therapy and/or more potent antilatency therapies may be needed.

In contrast to previous antiretroviral drugs, maraviroc does not need to cross the cell membrane, nor does not require intracellular processing in order to exert its activity. In addition, there is no cross-resistance between entry inhibitors and agents that act on intracellular targets.

Maraviroc has demonstrated potent antiviral activity against all CCR5-tropic HIV-1 viruses tested. Maraviroc could thus fulfil the requirements for an optimal candidate for treatment intensification in HIV-1 infected patients with a recent HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults (>=18 years old).
2. No previous antiretroviral therapy for more than 2 weeks.
3. HIV-1 infection documented in the past 6 months by a previous negative ELISA test, or a documented clinical acute seroconversion in the past 6 months.
4. CCR5-tropism confirmed at screening.
5. Voluntary written informed consent.

Exclusion Criteria:

1. Pregnancy or fertile women willing to be pregnant.
2. Active substance abuse or major psychiatric disease.
3. Presence of NRTI mutations in the screening genotype.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change at 48 weeks in the slope of decay of integrated and unintegrated viral DNA in PBMCs. | BL, W2, W4, W12, W24, W48

SECONDARY OUTCOMES:
Decay of residual HIV-1 replication under maraviroc intensification assessed by an ultrasensitive RT-PCR assay with a lower limit of quantification of 5 copies/mL. | BL, W2, W4, W8, W12, W24, W36, W48
Blips during the study (viral load >50 copies/mL, preceded and followed by determinations <50 copies/mL in previous and posterior controls). | From Baseline to W48
HIV-1 RNA below 50 copies/mL at 48 weeks. | W48
Change in the lymphocyte activation marker HLADR+CD38+ from baseline to week 48. | BL, W4, W12, W24, W48, W60, W72
Relationship between maraviroc and/or raltegravir plasma concentrations and change in the slope of decay of integrated viral DNA in PBMCs | W12, W24, W48
HIV-1 specific CTL responses | BL, W24, W48, W60, W72
Plasmatic inflammation biomarkers | BL, W2, W4, W12, W48, W60
RNA, DNA and viral p24 associated to cells in ileum biopsy and PBMC | W48
Lymphocyte activation marker HLADR+CD38+ in ileum biopsy and PBMC | W48
Fibrosis markers in ileum biopsy and PBMC | W48

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — LLuita contra la SIDA Foundation-HIV Unit; Josep Mª Llibre, MD,PhD, Principal Investigator — LLuita contra la SIDA Foundation-HIV Unit
Locations (2):
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona